CLINICAL TRIAL: NCT07255027
Title: Study on the Efficacy and Safety of Anesthesia-Induced Sleep Therapy for Refractory Insomnia: A Randomized Controlled Trial
Brief Title: Study on the Efficacy and Safety of Anesthesia-Induced Sleep Therapy for Refractory Insomnia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Inner Mongolia Autonomous Region Mental Health Center (Unknown)
Responsible Party: Principal Investigator, Yuming Peng, Deputy chief of Department of Anesthesiology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20250701
Record Dates: First submitted 2025-09-26; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Insomnia
Keywords: Anesthesia-Induced Sleep; Insomnia; Dexmedetomidine
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Active Comparator): Dexmedetomidine was administered intravenously once daily for three consecutive days, supplementing conventional oral drug therapy.
  Interventions: Drug: Dexmedetomidine and conventional oral drug
- Control group (Other): Patients only received conventional oral drug therapy.
  Interventions: Drug: Conventional oral drug therapy

INTERVENTIONS:
Drug: Dexmedetomidine and conventional oral drug — Dexmedetomidine was administered intravenously once daily for three consecutive days, supplementing conventional oral drug therapy. The dexmedetomidine was administered via a loading dose of 1.5 μg/kg intravenously over 15 minutes, with a subsequent continuous infusion at a maintenance dose of 0.5-0.7 μg/kg/h.
  Arms: Dexmedetomidine group
Drug: Conventional oral drug therapy — Patients only received conventional oral drug therapy.
  Arms: Control group

SUMMARY:
The incidence of refractory insomnia is rising annually, with traditional therapies offering limited efficacy. Anesthesia-Induced Sleep (AIS), involving anesthetic infusion like dexmedetomidine, is emerging. Its ability to mimic natural sleep architecture is unclear. Studies confirm AIS can shorten latency and improve sleep efficiency, but neuromodulatory mechanisms and long-term efficacy remain unclear with scarce follow-up data. This study used dexmedetomidine-based AIS under polysomnography to validate its induction of normal sleep architecture, evaluate long-term efficacy and safety, and explore mechanisms, aiming to provide a novel non-pharmacological intervention.

DETAILED DESCRIPTION:
The incidence of refractory insomnia has been rising annually, severely impacting patients' quality of life. Traditional pharmacological and physical therapies offer limited efficacy and struggle to achieve long-term relief. Anesthesia-Induced Sleep (AIS), an emerging treatment, typically involves intravenous infusion of anesthetic agents like dexmedetomidine to rapidly induce sleep. However, whether it can mimic natural sleep architecture remains unclear. Recent domestic and international studies have preliminarily confirmed that AIS can shorten latency and improve sleep efficiency. However, issues such as unclear neuromodulatory mechanisms and fluctuating long-term efficacy persist, and large-scale long-term follow-up data remain scarce. This study implemented dexmedetomidine-based AIS under polysomnographic monitoring to validate its ability to induce normal sleep architecture (e.g., restoring slow-wave sleep proportion) while evaluating long-term efficacy and safety. By quantifying sleep parameters and neural electrical activity, we explored potential mechanisms of AIS in reshaping sleep homeostasis. This research aims to provide a novel non-pharmacological intervention strategy for refractory insomnia and advance clinical translation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years meeting ICSD-3 diagnostic criteria for chronic insomnia.
* Persistent sleep disturbance (≥3 nights/week for ≥3 months).
* Significant daytime impairment (e.g., mood disturbance, cognitive decline).
* Treatment-refractory (failed prior pharmacotherapy/non-pharmacotherapy).
* No chronic obstructive pulmonary disease, moderate to severe sleep apnea syndrome, or atrioventricular block.
* Obtain written informed consent.

Exclusion Criteria:

* Participants with severe concomitant diseases affecting other organ systems.
* Moderate to severe obstructive sleep apnea (e.g., AHI ≥30 events/hour) or uncontrolled central sleep apnea.
* Pregnant, lactating, or planning pregnancy.
* History of alcoholism or drug dependence.
* Suicidal ideation or a severe psychiatric history (e.g., schizophrenia, unstable bipolar disorder).
* Participants with a prior allergic reaction to the study drug.
* Participants who have recently participated in other clinical studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of NREM-N3 sleep within total sleep time, as recorded by polysomnogram the night before discharge,an average of 7 days. | At the night before discharge,an average of 7 days.
  After the end of anesthesia-induced sleep therapy, the percentage of NREM-N3 recorded by polysomnogram within total sleep time at the night before discharge,an average of 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Peng, MD,Ph.D, Principal Investigator — Beijing Tiantan Hospital

IPD SHARING:
Plan to Share IPD: Undecided